CLINICAL TRIAL: NCT02034071
Title: A Dose Titration Study of Diazoxide Choline Controlled-Release Tablet (DCCR) in Patients With Prader-Willi Syndrome With a Double-Blind, Placebo-Controlled, Randomized Withdrawal Extension
Brief Title: Clinical Study of Diazoxide Choline Controlled-Release Tablet (DCCR) in Patients With Prader-Willi Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essentialis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC025
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCCR Open Label - DCCR Double Blind (Experimental): Patients are initiated on a DCCR dose of about 1.5 mg/kg (maximum starting dose of 145 mg) and are titrated every 14 days through 4 dose levels of DCCR. Patients will be up-titrated at each visit at the discretion of the investigator. Randomized to continue DCCR, at the same dose as they received on Day 69, in the Double-Blind, Placebo-Controlled, Randomized Withdrawal Extension
  Interventions: Drug: DCCR
- DCCR Open Label - Placebo Double Blind (Experimental): Patients are initiated on a DCCR dose of about 1.5 mg/kg (maximum starting dose of 145 mg) and are titrated every 14 days through 4 dose levels of DCCR. Patients will be up-titrated at each visit at the discretion of the investigator. Randomized to receive placebo equivalent to the DCCR dose received on Day 69 in the Double-Blind, Placebo-Controlled, Randomized Withdrawal Extension
  Interventions: Drug: DCCR; Drug: Placebo

INTERVENTIONS:
Drug: DCCR
  Other Names: Diazoxide Choline Controlled-Release Tablet
Drug: Placebo
  Arms: DCCR Open Label - Placebo Double Blind

SUMMARY:
• This is a single-center, open-label, single-arm study with a double-blind, placebo-controlled, randomized withdrawal extension. Patients are initiated on a DCCR dose of about 1.5 mg/kg (maximum starting dose of 145 mg) and are titrated every 14 days to about 2.4 mg/kg, 3.3 mg/kg, 4.2 mg/kg, and 5.1 mg/kg (maximum dose of 507.5 mg). These DCCR doses are equivalent to diazoxide doses of 1.03, 1.66, 2.28, 2.9, and 3.52 mg/kg. The administered dose will be as close to the mg/kg dosing as can be achieved by the available dose strengths of DCCR. Patients will be up-titrated at each visit at the discretion of the investigator. All patients will be continued in the double-blind, placebo-controlled, randomized withdrawal extension. Any patient who showed an increase in resting energy expenditure and/or a reduction in hyperphagia from Baseline through Day 55 or Day 69 will be designated a responder, whereas all others will be designated non-responders. Responders will be randomized in a 1:1 ratio either to continue on active treatment at the dose they were treated with on Day 69 or to the placebo equivalent of that dose for an additional 4 weeks. Non-responders will continue open label treatment during the extension.

ELIGIBILITY:
Inclusion Criteria:

* Children. adolescents and young adults with genetically confirmed Prader-Willi syndrome
* Ages at ≥ 10 years and ≤ 22 years
* Generally healthy as documented by the medical history, physical examination, vital sign assessments, 12-lead electrocardiogram (ECG), and clinical laboratory assessments
* BMI exceeds the 95th percentile of the age specific BMI value on the CDC BMI charts
* Fasting glucose ≤ 126 mg/dL
* HbA1c ≤ 6.5 %

Exclusion Criteria:

* Administration of investigational drugs within 1 month prior to Screening Visit
* Anticipated requirement for use of prohibited medications
* History of allergic reaction or significant intolerance to: diazoxide, thiazides or sulfonamides
* Anticipate transitions in their care from family home to group home or other similar potentially disruptive changes
* Congestive heart failure or known compromised cardiac reserve
* Any other clinically significant endocrine, cardiovascular, pulmonary, neurological, psychiatric, hepatic, gastrointestinal, hematological, renal, or dermatological disease interfering with the assessments of the investigational drug, according to the Investigator

Ages: 10 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Hyperphagia using hyperphagia questionnaire | Change from Day 69 through Day 97
Resting energy expenditure | Change from Day 69 through Day 97

OTHER OUTCOMES:
Weight | Percent Change from Baseline through Day 69
Weight | Percent Change from Day 69 through Day 97
Resting energy expenditure | Change from Baseline through Day 69
Hyperphagia using hyperphagia questionnaire | Change from Baseline through Day 69
Percent Body Fat | Change from Baseline through Day 69
Percent Body Fat | Change from Day 69 through Day 97
Lipids | Percent Change from Baseline through Day 69
  Percent change from Baseline through Day 69 for triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol, and non-HDL cholesterol
Lipids | Percent Change from Day 69 Through Day 97
  Percent change from Day 69 through Day 97 for triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol, and non-HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kimonis, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Orange, California, United States

REFERENCES:
- See also: Prader-Willi Syndrome Association USA — http://www.pwsausa.org/
- See also: Genetics Home Reference - Prader-Willi syndrome — http://ghr.nlm.nih.gov/condition/prader-willi-syndrome
- See also: Foundation for Prader-Willi Research - About Prader-Willi syndrome — http://www.fpwr.org/about-prader-willi-syndrome